CLINICAL TRIAL: NCT02613897
Title: A 16-wk, Uni-center, Randomized, Double-blind, Parallel, Phase 3b Trial to Evaluate Efficacy of Saxagliptin + Dapagliflozin vs.Dapagliflozin With Regard to EGP in T2DM With Insufficient Glycemic Control on Metformin+/-Sulfonylurea Therapy
Brief Title: ESR-15-11293 - Saxa/Dapa, Safety and Efficacy Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HSC20150742H
Record Dates: First submitted 2015-11-12; First posted 2015-11-25 (Estimated); Results first posted 2019-08-14 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-06

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — saxagliptin; dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- DAPA/SAXA (dapagliflozin plus saxagliptin) (Active Comparator): Dapagliflozin 10mg + Saxagliptin 5mg (plus standard of care treatment of metformin or metformin plus sulfonylurea).
  Interventions: Drug: Saxagliptin; Drug: Dapagliflozin
- DAPA (Dapagliflozin plus placebo) (Active Comparator): Dapagliflozin 10mg + Placebo (plus standard of care treatment of metformin or metformin plus sulfonylurea).
  Interventions: Drug: Dapagliflozin
- PCB (Placebo plus placebo) (Placebo Comparator): Placebo (for dapagliflozin) + placebo (for saxagliptin) (plus standard of care treatment of metformin or metformin plus sulfonylurea).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Saxagliptin — Saxagliptin (Onglyza™) is approved by the US FDA as an adjunct to diet and exercise to improve glycemic control in adults with T2DM. The 5 mg dose will be used for this study as it is the dose that is routinely used in the clinic. In addition, this dose is used in the pivotal studies in the saxagliptin/dapagliflozin clinical program.
  Other Names: Onglyza
  Arms: DAPA/SAXA (dapagliflozin plus saxagliptin)
Drug: Dapagliflozin — Dapagliflozin (Farxiga) is approved by the FDA as an adjunct to diet and exercise to improve glycemic control in adults with T2DM. Dapagliflozin (Farxiga) is also approved in the EU as an adjunct to diet and exercise to improve glycemic control in patients with T2DM for whom metformin use is considered inappropriate due to intolerance, and in combination with other glucose-lowering medicinal products when these, in combination with diet and exercise do not provide adequate glycemic control. The 10 mg dose was chosen for this study because it has been extensively studied in Phase 3 trials and has demonstrated a favorable benefit-risk profile. In addition, this dose is the most commonly used dose in most countries.
  Other Names: Farxiga
  Arms: DAPA (Dapagliflozin plus placebo); DAPA/SAXA (dapagliflozin plus saxagliptin)
Drug: Placebo — Placebo
  Arms: PCB (Placebo plus placebo)

SUMMARY:
This is a 16-week, single center, randomized, double-blind, active-controlled, parallel-group, Phase 3b efficacy and safety study of simultaneous administration of saxagliptin 5 mg plus dapagliflozin 10 mg once daily (QD) compared with dapagliflozin plus placebo for saxagliptin, and placebo for saxagliptin plus placebo for dapagliflozin in patients with Type 2 diabetes who have inadequate glycemic control on metformin or metformin/sulfonylurea.

DETAILED DESCRIPTION:
The study is intended to demonstrate complimentary action of saxagliptin/dapagliflozin added to metformin versus dapagliflozin added to metformin with regard to EGP.

Many medications are approved for the treatment of T2DM; however, the challenge of achieving and maintaining treatment goals within the current sequential therapy approach is linked to shortcomings of older classes of drugs. Metformin is in the biguanide drug class that acts to decrease hepatic glucose output and subsequently, decreases fasting hyperglycemia. Metformin, the oral first-line gold standard agent, is recommended as the initial pharmacological therapy because of its glycemic efficacy, weight neutrality, low risk of hypoglycemia, and beneficial cardiovascular (CV) profile. Current sequential add-on second and third line oral therapy includes oral drugs such as sulfonylureas (SUs) and thiazolidinediones (TZDs). These therapies and insulin are associated with increased risks for weight gain and hypoglycemia; therefore, caution is recommended when using combination therapy with other agents known to cause hypoglycemia. Hypoglycemia is a clinically important issue in optimizing treatment and there is emerging evidence that hypoglycemia is associated with negative CV outcomes. Efforts by patients to lose weight as part of a therapeutic lifestyle program are undermined by therapies that lead to weight gain. The majority of patients with T2DM are overweight or obese, and additional weight gain often results in reduced treatment efficacy.

Over the past few years, it has been widely recognized that the management approach for each T2DM patients' needs to be personalized based on his or her clinical characteristics (e.g., the likelihood of weight gain, risk for hypoglycemia, and lifestyle preferences [e.g., many patients may be reluctant to use injections]) (Inzucchi et al 2012). Based on data from the National Health and Nutrition Examination Survey in 2007 to 2010, HbA1c is not appropriately controlled in approximately one-third of patients using even less stringent targets (Ali et al 2013).

Because of the challenge to achieve glycemic control in patients with T2DM, the progressive nature of the disease, and the limitations of available oral and non-oral therapies, there is a significant medical need for oral combination treatment options and dual add-on therapy in patients with high baseline HbA1c. Expert groups have increasingly suggested making use of combination therapy early after diagnosis to improve glycemic control (Inzucchi et al 2012, Rodbard et al 2009). In a recent study, initiating triple therapy (pathophysiological-based approach) in patients with new onset T2DM versus metformin followed by sequential addition of SUs and basal insulin (treat-to-fail approach) demonstrated a more durable HbA1c reduction over 24 months and less hypoglycemia with initial triple therapy (Abdul-Ghani et al 2014). Initial combination therapy with saxagliptin and dapagliflozin added to metformin may have similar potential for durable glucose lowering in combination with low risk of hypoglycemia.

Treatment with saxagliptin and dapagliflozin, both individually and in combination with metformin, have demonstrated a favorable safety and tolerability profile. These drugs had a low propensity for hypoglycemia, therefore addressing a potential key concern when adding 2 glucose lowering agents simultaneously. These drugs have demonstrated weight neutrality (saxagliptin) or moderate weight reduction (dapagliflozin). Dapagliflozin has also been shown to cause a persistent reduction in HbA1c and weight after 2 years of therapy. Dapagliflozin was recently shown to increase EGP, which, in part, may be mediated by increased plasma glucagon (Merovci et al). In contrast, saxagliptin has been demonstrated to reduce glucagon levels, e.g., in response to a meal (Sjöstrand et al 2014) and vildagliptin, also a DPP-4 inhibitor, has been shown to inhibit EGP (Balas et al 2007).

A second-line oral dual add-on therapy with saxagliptin co-administered with dapagliflozin could be a new option, as part of a triple therapy combination that includes drugs with complementary mechanisms of action, opposing effects on plasma glucagon concentration, and possibly EGP, low risk of hypoglycemia, and the potential for moderate weight loss, providing a more effective and patient-friendly approach to the treatment of T2DM.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent prior to any study-specific procedures.
2. Is able to read, understand, and sign the Informed Consent Forms (ICFs) and, if applicable, an Authorization to Use and Disclose Protected Health Information form (consistent with Health Insurance Portability and Accountability Act of 1996 legislation), communicate with the Investigator, and understand and comply with protocol requirements, including the use of diary and glucose meter measurements.
3. Age = 18-70 years.
4. Has a diagnosis of T2DM.
5. Has HbA1c ≥7.5% and ≤11.0% obtained at Screening.
6. Treated with a stable dose of metformin ≥1000 mg/day or stable dose of metformin (≥ 1000 mg/day) plus sulfonylurea (glipizide, ≥ 5 mg/day; glyburide, ≥ 5 mg/day; glimepiride, ≥ 4 mg/day) for at least 8 weeks prior to Screening.
7. Has a BMI of 20 to 45 kg/m2 (inclusive) at Screening.
8. Is male, or is female, and meets all the following criteria:

   * Not pregnant or breastfeeding.
   * Negative pregnancy test result at Visit 1 (Screening).
   * Women of childbearing potential (WOCBP; [including perimenopausal women who have had a menstrual period within 1 year]) must practice and be willing to continue to practice appropriate birth control (defined as a method that results in a low failure rate, i.e., less than 1% per year, when used consistently and correctly, such as implants, injectables, hormonal contraceptives [pills, vaginal rings, or patches], some intrauterine contraceptive devices [levonorgestrel-releasing or copper-T], tubal ligation or occlusion, or a vasectomized partner) during the entire duration of the study. As applicable, all methods must be in effect prior to receiving the first dose of study medication.

Exclusion Criteria:

Target Disease Exceptions

1. Clinically diagnosed with Type I diabetes .
2. History of diabetic ketoacidosis, hyperosmolar nonketotic coma, or corticosteroid induced Type 2 diabetes.

   Medical History and Concurrent Diseases
3. History of bariatric surgery or lap-band surgery, or either procedure is planned during the time period of the study.
4. History of any unstable endocrine, psychiatric, rapidly progressing, or unstable renal disease, or rheumatic disorder, as judged by the Investigator.
5. Patients who, in the judgment of the Investigator, may be at risk for dehydration or volume depletion that may affect the patient's safety and/or the interpretation of efficacy or safety data.
6. Has evidence of current abuse of drugs or alcohol or a history of abuse within the past 52 weeks that, in the Investigator's opinion, would cause the individual to be noncompliant.

   Cardiovascular Conditions
7. Cardiovascular disease within 3 months of Screening (i.e., MI, cardiac surgery, revascularization, unstable angina, stroke, transient ischemic attack, or arrhythmia).
8. Presence or history of severe congestive heart failure (New York Heart Association Class III and IV [CCNYHA 1994]), unstable or acute congestive heart failure, and/or known left ventricular ejection fraction of ≤40%.

   Note: Eligible patients with congestive heart failure, especially those who are on diuretic therapy, should have careful monitoring of their volume status throughout the study.

   Kidney Conditions
9. Estimated (eGFR) <60±5 mL/min/1.73 m2 or a measured serum creatinine of >1.4 mg/dL for female patients and >1.5 mg/dL for male patients. If the serum creatinine is ≤ 1.4 (female) or ≤ 1.5 (male) and the eGFR is ≥ 60±5 ml/min/1.73m2, the subject is eligible to participate in the study.
10. Congenital renal glucosuria. Hepatic Conditions
11. Significant hepatic disease, including, but not limited to, severe hepatic insufficiency and/or significant abnormal liver function defined as aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) of >3x upper limit of normal (ULN).
12. Serum total bilirubin (TB) >2 mg/dL.
13. History of, or currently have, acute or chronic pancreatitis or have triglyceride concentrations ≥500 mg/dL at Visit 1 (Screening).
14. Suspicion that the patient is infected with an infectious substance according to World Health Organization risk categories A and B (see Appendix C).
15. Known severe hepatic disease, including chronic active hepatitis.
16. Positive serologic evidence of current infectious liver disease, including patients positive for hepatitis B viral antibody IgM, hepatitis B surface antigen, and hepatitis C virus antibody.

    Hematological/Oncological Conditions
17. Malignancy within 5 years of Visit 1 (Screening), with the exception of treated in situ basal cell or squamous cell carcinoma of the skin.
18. Hematocrit of <34% for both males and females. Prohibited Medications
19. Administration of any antihyperglycemic therapy, other than metformin or metformin/sulfonylurea, for more than 14 days (consecutive or not) during the 12 weeks prior to Visit 1 (Screening) and during the study unless per protocol for rescue.
20. Current treatment with potent cytochrome P450 3A4/5 inhibitors (e.g., atazanavir, clarithromycin, indinavir, itraconazole, nefazodone, nelfinavir, ritonavir, saquinavir, and telithromycin).
21. Administration of any other investigational drug or participation in any interventional clinical studies 30 days prior to Visit 1 (Screening).
22. Treatment with systemic corticosteroids for the last 3 months prior to Visit 1 (Screening).
23. Prescription or over-the-counter weight loss medications within 3 months prior to Visit 1 (Screening).

    Other
24. Patients with abnormal thyroid stimulating hormone (TSH) or free thyroxine (T4) values at Visit 1 (Screening) will be excluded.
25. Has a clinically significant medical condition that could potentially affect study participation and/or personal well-being, as judged by the Investigator.
26. Has clinically significant abnormal laboratory test values (clinical chemistry, hematology, and urinalysis) as judged by the Investigator at Visit 1 (Screening).
27. Has known contraindications, allergies, or hypersensitivities to any study medication or excipient as outlined in the IBs or local package inserts for saxagliptin and dapagliflozin.
28. Has a contraindication to metformin use, including known metabolic or lactic acidosis, or any condition associated with hypoperfusion, hypoxemia, dehydration, or sepsis.
29. Is currently pregnant (confirmed with positive pregnancy test) or breast feeding.
30. Is on a commercial weight loss program with ongoing weight loss more than 5% over the last 3 months prior to Visit 1 (Screening), or is on an intensive exercise program.
31. Involvement in the planning and/or conduct of the study (applies to both the study sponsor staff and/or staff at the study site).
32. Patient with any condition that, in the judgment of the Investigator, may render the patient unable to complete the study or which may pose a significant risk to the patient or patient suspected or with confirmed poor protocol or medication compliance.
33. Previous randomization in the present study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2016-01; Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eugenio Cersosimo, MD, Principal Investigator — The University of Texas Health Science Center at San Antonio; Ralph A DeFronzo, MD, Study Director — The University of Texas Health Science Center at San Antonio
Locations (1):
- The University of Texas Health Science Center at San Antonio, San Antonio, Texas, United States

REFERENCES:
- [Background] Rodbard HW, Blonde L, Braithwaite SS, Brett EM, Cobin RH, Handelsman Y, Hellman R, Jellinger PS, Jovanovic LG, Levy P, Mechanick JI, Zangeneh F; AACE Diabetes Mellitus Clinical Practice Guidelines Task Force. American Association of Clinical Endocrinologists medical guidelines for clinical practice for the management of diabetes mellitus. Endocr Pract. 2007 May-Jun;13 Suppl 1:1-68. doi: 10.4158/EP.13.S1.1. No abstract available. PMID 17613449
- [Background] Abdul-Ghani MA, Norton L, Defronzo RA. Role of sodium-glucose cotransporter 2 (SGLT 2) inhibitors in the treatment of type 2 diabetes. Endocr Rev. 2011 Aug;32(4):515-31. doi: 10.1210/er.2010-0029. Epub 2011 May 23. PMID 21606218
- [Background] Abdul-Ghani MA, Puckett C, Triplitt C, Maggs D, Adams J, Cersosimo E, DeFronzo RA. Initial combination therapy with metformin, pioglitazone and exenatide is more effective than sequential add-on therapy in subjects with new-onset diabetes. Results from the Efficacy and Durability of Initial Combination Therapy for Type 2 Diabetes (EDICT): a randomized trial. Diabetes Obes Metab. 2015 Mar;17(3):268-75. doi: 10.1111/dom.12417. Epub 2015 Jan 7. PMID 25425451
- [Background] Ali MK, Bullard KM, Gregg EW. Achievement of goals in U.S. Diabetes Care, 1999-2010. N Engl J Med. 2013 Jul 18;369(3):287-8. doi: 10.1056/NEJMc1306652. No abstract available. PMID 23863067
- [Background] Balas B, Baig MR, Watson C, Dunning BE, Ligueros-Saylan M, Wang Y, He YL, Darland C, Holst JJ, Deacon CF, Cusi K, Mari A, Foley JE, DeFronzo RA. The dipeptidyl peptidase IV inhibitor vildagliptin suppresses endogenous glucose production and enhances islet function after single-dose administration in type 2 diabetic patients. J Clin Endocrinol Metab. 2007 Apr;92(4):1249-55. doi: 10.1210/jc.2006-1882. Epub 2007 Jan 23. PMID 17244786
- [Background] The Criteria Committee of the New York Heart Association. Nomenclature and Criteria for Diagnosis of Diseases of the Heart and Great Vessels. (9th ed.). Boston: Little, Brown & Co. 1994; 253-256.
- [Background] Centers for Disease Control and Prevention (CDC). Prevalence of overweight and obesity among adults with diagnosed diabetes--United States, 1988-1994 and 1999-2002. MMWR Morb Mortal Wkly Rep. 2004 Nov 19;53(45):1066-8. PMID 15549021
- [Background] CHMP 2009 European Medicines Agency (EMA) Committee for Medicinal Products for Human Use (CHMP). Guideline on Clinical Development of Fixed Combination Medicinal Products. CHMP/EWP/240/95 Rev. 1. Available at: http://www.ema.europa.eu/docs/en_GB/document_library/Scientific_guideline/2009/09/WC500003686.pdf. Published 19 February 2009. Accessed 19 June 2014.
- [Background] CHMP 2012 European Medicines Agency (EMA) Committee for Medicinal Products for Human Use (CHMP). Guideline on clinical investigation of medicinal products in the treatment or prevention of diabetes mellitus. CPMP/EWP/1080/00 Rev. 1. Available at: http://www.ema.europa.eu/docs/en_GB/document_library/Scientific_guideline/2012/06/WC500129256.pdf. Published 14 May 2012. Accessed 19 June 2014.
- [Background] Defronzo RA. Banting Lecture. From the triumvirate to the ominous octet: a new paradigm for the treatment of type 2 diabetes mellitus. Diabetes. 2009 Apr;58(4):773-95. doi: 10.2337/db09-9028. No abstract available. PMID 19336687
- [Background] Del Prato S, Barnett AH, Huisman H, Neubacher D, Woerle HJ, Dugi KA. Effect of linagliptin monotherapy on glycaemic control and markers of beta-cell function in patients with inadequately controlled type 2 diabetes: a randomized controlled trial. Diabetes Obes Metab. 2011 Mar;13(3):258-67. doi: 10.1111/j.1463-1326.2010.01350.x. PMID 21205122
- [Background] Dicker D. DPP-4 inhibitors: impact on glycemic control and cardiovascular risk factors. Diabetes Care. 2011 May;34 Suppl 2(Suppl 2):S276-8. doi: 10.2337/dc11-s229. No abstract available. PMID 21525468
- [Background] Diabetes Control and Complications Trial Research Group; Nathan DM, Genuth S, Lachin J, Cleary P, Crofford O, Davis M, Rand L, Siebert C. The effect of intensive treatment of diabetes on the development and progression of long-term complications in insulin-dependent diabetes mellitus. N Engl J Med. 1993 Sep 30;329(14):977-86. doi: 10.1056/NEJM199309303291401. PMID 8366922
- [Background] Ferrannini E, Bjorkman O, Reichard GA Jr, Pilo A, Olsson M, Wahren J, DeFronzo RA. The disposal of an oral glucose load in healthy subjects. A quantitative study. Diabetes. 1985 Jun;34(6):580-8. doi: 10.2337/diab.34.6.580. PMID 3891471
- [Background] Goke B, Hershon K, Kerr D, Calle Pascual A, Schweizer A, Foley J, Shao Q, Dejager S. Efficacy and safety of vildagliptin monotherapy during 2-year treatment of drug-naive patients with type 2 diabetes: comparison with metformin. Horm Metab Res. 2008 Dec;40(12):892-5. doi: 10.1055/s-0028-1082334. Epub 2008 Aug 22. PMID 18726829
- [Background] Gomis R, Espadero RM, Jones R, Woerle HJ, Dugi KA. Efficacy and safety of initial combination therapy with linagliptin and pioglitazone in patients with inadequately controlled type 2 diabetes: a randomized, double-blind, placebo-controlled study. Diabetes Obes Metab. 2011 Jul;13(7):653-61. doi: 10.1111/j.1463-1326.2011.01391.x. PMID 21410628
- [Background] Hansen L, Iqbal N, Ekholm E, Cook W, Hirshberg B. Postprandial dynamics of plasma glucose, insulin, and glucagon in patients with type 2 diabetes treated with saxagliptin plus dapagliflozin add-on to metformin therapy. Endocr Pract. 2014 Nov;20(11):1187-97. doi: 10.4158/EP14489.OR. PMID 25370334
- [Background] Hoerger TJ, Segel JE, Gregg EW, Saaddine JB. Is glycemic control improving in U.S. adults? Diabetes Care. 2008 Jan;31(1):81-6. doi: 10.2337/dc07-1572. Epub 2007 Oct 12. PMID 17934153
- [Background] Inzucchi SE, Bergenstal RM, Buse JB, Diamant M, Ferrannini E, Nauck M, Peters AL, Tsapas A, Wender R, Matthews DR; American Diabetes Association (ADA); European Association for the Study of Diabetes (EASD). Management of hyperglycemia in type 2 diabetes: a patient-centered approach: position statement of the American Diabetes Association (ADA) and the European Association for the Study of Diabetes (EASD). Diabetes Care. 2012 Jun;35(6):1364-79. doi: 10.2337/dc12-0413. Epub 2012 Apr 19. No abstract available. PMID 22517736
- [Background] Jani R, Molina M, Matsuda M, Balas B, Chavez A, DeFronzo RA, Abdul-Ghani M. Decreased non-insulin-dependent glucose clearance contributes to the rise in fasting plasma glucose in the nondiabetic range. Diabetes Care. 2008 Feb;31(2):311-5. doi: 10.2337/dc07-1593. Epub 2007 Nov 13. PMID 18000182
- [Background] Klein S, Sheard NF, Pi-Sunyer X, Daly A, Wylie-Rosett J, Kulkarni K, Clark NG; American Diabetes Association; North American Association for the Study of Obesity; American Society for Clinical Nutrition. Weight management through lifestyle modification for the prevention and management of type 2 diabetes: rationale and strategies: a statement of the American Diabetes Association, the North American Association for the Study of Obesity, and the American Society for Clinical Nutrition. Diabetes Care. 2004 Aug;27(8):2067-73. doi: 10.2337/diacare.27.8.2067. No abstract available. PMID 15277443
- [Background] Komoroski B, Vachharajani N, Boulton D, Kornhauser D, Geraldes M, Li L, Pfister M. Dapagliflozin, a novel SGLT2 inhibitor, induces dose-dependent glucosuria in healthy subjects. Clin Pharmacol Ther. 2009 May;85(5):520-6. doi: 10.1038/clpt.2008.251. Epub 2009 Jan 7. PMID 19129748
- [Background] Merovci A, Solis-Herrera C, Daniele G, Eldor R, Fiorentino TV, Tripathy D, Xiong J, Perez Z, Norton L, Abdul-Ghani MA, DeFronzo RA. Dapagliflozin improves muscle insulin sensitivity but enhances endogenous glucose production. J Clin Invest. 2014 Feb;124(2):509-14. doi: 10.1172/JCI70704. Epub 2014 Jan 27. PMID 24463448
- [Background] Nathan DM, Buse JB, Davidson MB, Ferrannini E, Holman RR, Sherwin R, Zinman B. Management of hyperglycaemia in type 2 diabetes mellitus: a consensus algorithm for the initiation and adjustment of therapy. Update regarding the thiazolidinediones. Diabetologia. 2008 Jan;51(1):8-11. doi: 10.1007/s00125-007-0873-z. No abstract available. PMID 18026926
- [Background] NHLBI 1998 National Heart, Lung, and Blood Institute (NHLBI) Clinical Guidelines on the Identification, Evaluation, and Treatment of Overweight and Obesity in Adults. NIH publication No. 98 4083. Available at: http://www.nhlbi.nih.gov/guidelines/obesity/ob_home.htm. Published September 1998. Accessed 19 June 2014.
- [Background] Owens DR, Swallow R, Dugi KA, Woerle HJ. Efficacy and safety of linagliptin in persons with type 2 diabetes inadequately controlled by a combination of metformin and sulphonylurea: a 24-week randomized study. Diabet Med. 2011 Nov;28(11):1352-61. doi: 10.1111/j.1464-5491.2011.03387.x. PMID 21781152
- [Background] Qaseem A, Vijan S, Snow V, Cross JT, Weiss KB, Owens DK; Clinical Efficacy Assessment Subcommittee of the American College of Physicians. Glycemic control and type 2 diabetes mellitus: the optimal hemoglobin A1c targets. A guidance statement from the American College of Physicians. Ann Intern Med. 2007 Sep 18;147(6):417-22. doi: 10.7326/0003-4819-147-6-200709180-00012. PMID 17876024
- [Background] Rodbard HW, Jellinger PS, Davidson JA, Einhorn D, Garber AJ, Grunberger G, Handelsman Y, Horton ES, Lebovitz H, Levy P, Moghissi ES, Schwartz SS. Statement by an American Association of Clinical Endocrinologists/American College of Endocrinology consensus panel on type 2 diabetes mellitus: an algorithm for glycemic control. Endocr Pract. 2009 Sep-Oct;15(6):540-59. doi: 10.4158/EP.15.6.540. PMID 19858063
- [Background] Scirica BM, Bhatt DL, Braunwald E, Steg PG, Davidson J, Hirshberg B, Ohman P, Frederich R, Wiviott SD, Hoffman EB, Cavender MA, Udell JA, Desai NR, Mosenzon O, McGuire DK, Ray KK, Leiter LA, Raz I; SAVOR-TIMI 53 Steering Committee and Investigators. Saxagliptin and cardiovascular outcomes in patients with type 2 diabetes mellitus. N Engl J Med. 2013 Oct 3;369(14):1317-26. doi: 10.1056/NEJMoa1307684. Epub 2013 Sep 2. PMID 23992601
- [Background] Seaquist ER, Anderson J, Childs B, Cryer P, Dagogo-Jack S, Fish L, Heller SR, Rodriguez H, Rosenzweig J, Vigersky R. Hypoglycemia and diabetes: a report of a workgroup of the American Diabetes Association and the Endocrine Society. Diabetes Care. 2013 May;36(5):1384-95. doi: 10.2337/dc12-2480. Epub 2013 Apr 15. PMID 23589542
- [Background] Sjostrand M, Iqbal N, Lu J, Hirshberg B. Saxagliptin improves glycemic control by modulating postprandial glucagon and C-peptide levels in Chinese patients with type 2 diabetes. Diabetes Res Clin Pract. 2014 Aug;105(2):185-91. doi: 10.1016/j.diabres.2014.05.006. Epub 2014 May 29. PMID 24947443
- [Background] Taskinen MR, Rosenstock J, Tamminen I, Kubiak R, Patel S, Dugi KA, Woerle HJ. Safety and efficacy of linagliptin as add-on therapy to metformin in patients with type 2 diabetes: a randomized, double-blind, placebo-controlled study. Diabetes Obes Metab. 2011 Jan;13(1):65-74. doi: 10.1111/j.1463-1326.2010.01326.x. PMID 21114605
- [Background] Intensive blood-glucose control with sulphonylureas or insulin compared with conventional treatment and risk of complications in patients with type 2 diabetes (UKPDS 33). UK Prospective Diabetes Study (UKPDS) Group. Lancet. 1998 Sep 12;352(9131):837-53. PMID 9742976
- [Background] Effect of intensive blood-glucose control with metformin on complications in overweight patients with type 2 diabetes (UKPDS 34). UK Prospective Diabetes Study (UKPDS) Group. Lancet. 1998 Sep 12;352(9131):854-65. PMID 9742977
- [Derived] Qin Y, Adams J, Solis-Herrera C, Triplitt C, DeFronzo R, Cersosimo E. Clinical Parameters, Fuel Oxidation, and Glucose Kinetics in Patients With Type 2 Diabetes Treated With Dapagliflozin Plus Saxagliptin. Diabetes Care. 2020 Oct;43(10):2519-2527. doi: 10.2337/dc19-1993. Epub 2020 Jul 21. PMID 32694214

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | DAPA/SAXA (Dapagliflozin Plus Saxagliptin) | DAPA (Dapagliflozin Plus Placebo) | PCB (Placebo Plus Placebo)
Started | 22 | 22 | 12
Completed | 22 | 22 | 12
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Dapa/Saxa: Subjects with type 2 diabetes were enrolled into this study and received the intervention of Dapagliflozin plus Saxa
- Dapa/Placebo: Subjects with type 2 diabetes were enrolled into this study and received the intervention of Dapagliflozin plus placebo
- Placebo/Placebo: Subjects with type 2 diabetes were enrolled into this study and received the intervention of placebo plus placebo
- Total: Total of all reporting groups
Arm/Group | Dapa/Saxa | Dapa/Placebo | Placebo/Placebo | Total
Number analyzed (Participants) | 22 | 22 | 12 | 56
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52 (2) | 52 (2) | 52 (2) | 52 (2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 14 | 2 | 29
  Male | 9 | 8 | 10 | 27
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic | 18 | 18 | 9 | 45
  White | 2 | 2 | 1 | 5
  Black | 2 | 0 | 2 | 4
  Asian | 0 | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 22 | 22 | 12 | 56

OUTCOME MEASURES:

1. Primary Outcome: Change in Endogenous Glucose Production (EGP)
Description: All subjects received a Double-Tracer Oral Glucose Tolerance Test (OGTT) with 75g of glucose containing 14C-glucose together with intravenous primed-continuous infusion of 3(3H)-glucose for 240 minutes, at baseline (prior to) and after 16 weeks of therapy. Blood and urine samples were obtained during the OGTT to determine EGP.
Time Frame: Baseline and 16 weeks
Measure: Mean (Standard Error); unit: mg/kg*min
Arm/Group | DAPA/SAXA (Dapagliflozin Plus Saxagliptin) | DAPA (Dapagliflozin Plus Placebo) | PCB (Placebo Plus Placebo)
Number analyzed (Participants) | 22 | 22 | 12
mg/kg*min
  Baseline Measurement | 2.45 (0.05) | 2.56 (0.04) | 1.95 (0.05)
  16 weeks | 2.4 (0.02) | 2.8 (0.01) | 2.15 (0.02)

2. Secondary Outcome: Change in Body Weight
Description: Change in body weight from baseline to 16 weeks
Time Frame: Baseline to 16 weeks
Measure: Mean (Standard Deviation); unit: Kg
Arm/Group | DAPA/SAXA (Dapagliflozin Plus Saxagliptin) | DAPA (Dapagliflozin Plus Placebo) | PCB (Placebo Plus Placebo)
Number analyzed (Participants) | 22 | 22 | 12
Kg | -2.28 (0.67) | -1.76 (0.88) | 0.26 (0.7)

3. Secondary Outcome: Change in BMI
Description: Change in BMI (body mass index) from study start to 16 weeks
Time Frame: Change from baseline to 16 weeks
Measure: Mean (Standard Deviation); unit: Kg/m^2
Arm/Group | DAPA/SAXA (Dapagliflozin Plus Saxagliptin) | DAPA (Dapagliflozin Plus Placebo) | PCB (Placebo Plus Placebo)
Number analyzed (Participants) | 22 | 22 | 12
Kg/m^2 | -0.8 (0.24) | -0.66 (0.33) | 0.16 (0.24)

4. Secondary Outcome: HBA1c
Description: Change in blood glucose level measured over a 3 month period from study start to 16 weeks
Time Frame: Change from baseline to 16 weeks
Measure: Mean (Standard Deviation); unit: percentage change in blood glucose level
Arm/Group | DAPA/SAXA (Dapagliflozin Plus Saxagliptin) | DAPA (Dapagliflozin Plus Placebo) | PCB (Placebo Plus Placebo)
Number analyzed (Participants) | 22 | 22 | 12
percentage change in blood glucose level | -1.67 (0.35) | -1.46 (0.22) | 0.44 (0.36)

5. Secondary Outcome: Mean Oral Glucose Tolerance Test (OGTT)
Description: Measure of change in OGTT from study start to 16 weeks
Time Frame: Change from baseline to 16 weeks
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | DAPA/SAXA (Dapagliflozin Plus Saxagliptin) | DAPA (Dapagliflozin Plus Placebo) | PCB (Placebo Plus Placebo)
Number analyzed (Participants) | 22 | 22 | 12
mg/dl | -49.62 (9.03) | -44.24 (7.76) | 20.26 (9.25)

6. Secondary Outcome: Change in Lipid Oxidation
Description: Change in lipid oxidation percentage from baseline to 16 weeks
Time Frame: Change from baseline to 16 weeks
Measure: Mean (Standard Deviation); unit: percentage of oxidation
Arm/Group | DAPA/SAXA (Dapagliflozin Plus Saxagliptin) | DAPA (Dapagliflozin Plus Placebo) | PCB (Placebo Plus Placebo)
Number analyzed (Participants) | 22 | 22 | 12
percentage of oxidation | -11.87 (2.52) | 22.02 (2.81) | -6.69 (4.95)

7. Secondary Outcome: Change in Glucose Oxidation
Description: Change in percentage of glucose oxidation from study start to 16 weeks
Time Frame: Change from baseline to 16 weeks
Measure: Mean (Standard Deviation); unit: percentage of oxidation
Arm/Group | DAPA/SAXA (Dapagliflozin Plus Saxagliptin) | DAPA (Dapagliflozin Plus Placebo) | PCB (Placebo Plus Placebo)
Number analyzed (Participants) | 22 | 22 | 12
percentage of oxidation | -22.07 (2.22) | -46.54 (2.79) | 4.65 (4.89)

8. Secondary Outcome: Change in Fasting Plasma Glucagon (FPG)
Description: A measure of the change in fasting plasma glucagon from study start to 16 weeks
Time Frame: Change from baseline to 16 weeks
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | DAPA/SAXA (Dapagliflozin Plus Saxagliptin) | DAPA (Dapagliflozin Plus Placebo) | PCB (Placebo Plus Placebo)
Number analyzed (Participants) | 22 | 22 | 12
mg/dl | -28.52 (5.74) | 26.89 (5.2) | 6.88 (5.09)

9. Secondary Outcome: Change in Free Fatty Acids (FFA)
Description: Measure of change in Free Fatty Acids from study start to 16 weeks
Time Frame: Change from baseline to 16 weeks
Measure: Mean (Standard Deviation); unit: mEq/L
Arm/Group | DAPA/SAXA (Dapagliflozin Plus Saxagliptin) | DAPA (Dapagliflozin Plus Placebo) | PCB (Placebo Plus Placebo)
Number analyzed (Participants) | 22 | 22 | 12
mEq/L | -0.06 (0.01) | -0.01 (0.02) | 0.00 (0.7)

ADVERSE EVENTS:
Time Frame: Adverse events were captured from baseline to 16 weeks
Arm/Group | DAPA/SAXA (Dapagliflozin Plus Saxagliptin) | DAPA (Dapagliflozin Plus Placebo) | PCB (Placebo Plus Placebo)
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/22 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22 | 0/12
Other Adverse Events (participants affected / at risk) | 11/22 | 9/22 | 3/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DAPA/SAXA (Dapagliflozin Plus Saxagliptin) (N=22) | DAPA (Dapagliflozin Plus Placebo) (N=22) | PCB (Placebo Plus Placebo) (N=12)
Increased urinary frequency (Renal and urinary disorders) | 3 (3) | 3 (3) | 1 (1)
Vaginal Itching (Reproductive system and breast disorders) | 2 (2) | 2 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Light headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dry Mouth (Gastrointestinal disorders) | 2 (2) | 2 (2) | 1 (1)
Urinary Tract Infection (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-30): https://cdn.clinicaltrials.gov/large-docs/97/NCT02613897/Prot_SAP_000.pdf